CLINICAL TRIAL: NCT05592587
Title: Evaluating Acceptance and Efficacy of an Eye Massage Device in Reducing Pain and Anxiety During Dental Anesthesia in Children.
Brief Title: Pain and Anxiety Reduction Using a Vibrating Eye Massage Device With Relaxing Nature Sounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Pedo-04-2022
Record Dates: First submitted 2022-09-17; First posted 2022-10-24 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Behavior, Child; Dental Anxiety; Anesthesia, Local
Keywords: Eye massage device; Vibratory stimulation; Nature sounds; Distraction
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Distraction using eye massage device producing both vibrations and nature sounds. (Experimental)
  Interventions: Behavioral: Evaluation of the effectiveness of eye massage device producing both vibrations and nature sounds distraction in the management of anxious pediatric patients during inferior alveolar nerve.
- Distraction using eye massage device producing vibratory stimulations only. (Experimental)
  Interventions: Behavioral: Evaluation of the effectiveness of eye massage device producing vibratory stimulations distraction in the management of anxious pediatric patients during inferior alveolar nerve.
- Using basic behavior guidance techniques and without using any type of distraction aids. (Other)
  Interventions: Behavioral: Evaluation of the effectiveness of basic behavior guidance techniques without using any type of distraction aids in the management of anxious pediatric patients during inferior alveolar nerve.

INTERVENTIONS:
Behavioral: Evaluation of the effectiveness of eye massage device producing both vibrations and nature sounds distraction in the management of anxious pediatric patients during inferior alveolar nerve. — The child will be provided inferior alveolar nerve during eye massage device producing both vibrations and nature sounds. Children will be assessed by using a combination of measures: Wong-Baker faces and the Children's Fear Scale (self-report), heart pulse rate and blood pressure (physiological), and behavior (using Anxiety levels using Face - Legs - Activity - Cry - Consolability "FLACC" scale "external evaluator"). Acceptance will be measured using a two-point Likert scale
  Arms: Distraction using eye massage device producing both vibrations and nature sounds.
Behavioral: Evaluation of the effectiveness of eye massage device producing vibratory stimulations distraction in the management of anxious pediatric patients during inferior alveolar nerve. — The child will be provided inferior alveolar nerve during eye massage device producing vibratory stimulations. Children will be assessed by using a combination of measures: Wong-Baker faces and the Children's Fear Scale (self-report), heart pulse rate and blood pressure (physiological), and behavior (using Anxiety levels using Face - Legs - Activity - Cry - Consolability "FLACC" scale "external evaluator"). Acceptance will be measured using a two-point Likert scale
  Arms: Distraction using eye massage device producing vibratory stimulations only.
Behavioral: Evaluation of the effectiveness of basic behavior guidance techniques without using any type of distraction aids in the management of anxious pediatric patients during inferior alveolar nerve. — The child will be provided inferior alveolar nerve during eye massage device producing vibratory stimulations. Children will be assessed by using a combination of measures: Wong-Baker faces and the Children's Fear Scale (self-report), heart pulse rate and blood pressure (physiological), and behavior (using Anxiety levels using Face - Legs - Activity - Cry - Consolability "FLACC" scale "external evaluator"). Acceptance will be measured using a two-point Likert scale
  Arms: Using basic behavior guidance techniques and without using any type of distraction aids.

SUMMARY:
This study aims to evaluate the effectiveness and acceptance of an eye massage device that produces nature sounds and vibratory stimulations in the management of anxious pediatric patients during inferior alveolar nerve block

Group A (Control group): inferior alveolar nerve block will be administrated with basic behavior guidance techniques and without distraction aids.

Group B: inferior alveolar nerve block will be administrated with the usage of the eye massage device producing both vibrations and nature sounds

Group C: inferior alveolar nerve block will be administrated with the eye massage device producing vibratory stimulations only.

All of the children who experienced an inferior alveolar block with/without distraction will be assessed by using a combination of measures: Wong-Baker faces and the Children's Fear Scale (self-report), heart pulse rate and blood pressure (physiological), and behavior (using Anxiety levels using Face - Legs - Activity - Cry - Consolability "FLACC" scale "external evaluator") Acceptance will be measured using a two-point Likert scale.

DETAILED DESCRIPTION:
This study will evaluate the effectiveness and acceptance of a distraction aid that produces both vibratory and natural sound stimulations. pain and anxiety will be assessed during inferior alveolar nerve block using four behavioral scales, Wong-Baker pain scale and Children's Fear Scale (self-report), pulse rate and blood pressure (physiological), and behavior (using FLACC behavior rating scale "external evaluator".

Heart pulse rate measurement will be recorded firstly when the patient is seated comfortably on the dental chair, during anesthesia, and finally, after the procedure is done and the child patients will be asked to choose a face that describes their status from one of both Wong Baker faces scale and Children's Fear Scale.

Blood pressure will be recorded before, during, and after anesthesia. Body responses of all child patients will be recorded during the whole procedure and then will be evaluated by an external evaluator to determine the children's behavioral score according to the FLACC scale.

ELIGIBILITY:
Inclusion Criteria:

1. age between 7 and 9 years.
2. no previous dental experience.
3. definitely positive or positive ratings of Frank scale.
4. Need of IAN block for any dental treatment.

Exclusion Criteria:

1. previous dental experience
2. systematic or mental disorders.
3. definitely negative or negative ratings of Frankel scale
4. Any contraindication for regional anesthesia

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Pain levels | 5 minutes following the inferior alveolar nerve block injection.
  Pain levels will be measured by using a self-reported simplified Wong-Baker faces pain scale:
  0 no Hurt - 1 Hurts little Bit - 2 Hurts little More - 3 Hurts Even More - 4 Hurts Whole Lot - 5 Hurts Worst
Anxiety levels | 1 minute during inferior alveolar nerve block administration.
  This will be evaluated using the Face-Legs-Activity-Cry-Consolability (FLACC) scale (0 low anxiety and pain level - 10 high anxiety and pain level).
Anxiety levels | five minutes following the inferior alveolar nerve block injection
  This will be evaluated using Children's Fear Scale (0 indicating 'no anxiety' and 4 indicating 'extreme anxiety').

SECONDARY OUTCOMES:
Pulse rate | (1) five minutes after the patient is seated comfortably on the dental chair, (2) five minutes following the injection of the anesthetic drug
  Pulse rate (the number of times your heart beats each minute bpm will be evaluated using Finger Pulse Oximeter.
Blood pressure | (1) five minutes after the patient is seated comfortably on the dental chair, (2) five minutes following the injection of the anesthetic drug
  Blood pressure (millimeters of mercury mmHg) will be evaluated using a Wrist Digital Blood Pressure Monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Dajma Abed, DDs, Principal Investigator — Damascus University; Nada G Bshara, Phd, Study Director — Damascus University
Locations (1):
- Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crego A, Carrillo-Diaz M, Armfield JM, Romero M. Dental fear and expected effectiveness of destructive coping as predictors of children's uncooperative intentions in dental settings. Int J Paediatr Dent. 2015 May;25(3):191-8. doi: 10.1111/ipd.12126. Epub 2014 Jul 22. PMID 25047094
- [Background] Attar RH, Baghdadi ZD. Comparative efficacy of active and passive distraction during restorative treatment in children using an iPad versus audiovisual eyeglasses: a randomised controlled trial. Eur Arch Paediatr Dent. 2015 Feb;16(1):1-8. doi: 10.1007/s40368-014-0136-x. Epub 2014 Nov 22. PMID 25416522
- [Background] Buxton RT, Pearson AL, Allou C, Fristrup K, Wittemyer G. A synthesis of health benefits of natural sounds and their distribution in national parks. Proc Natl Acad Sci U S A. 2021 Apr 6;118(14):e2013097118. doi: 10.1073/pnas.2013097118. PMID 33753555
- [Background] Canbulat N, Ayhan F, Inal S. Effectiveness of external cold and vibration for procedural pain relief during peripheral intravenous cannulation in pediatric patients. Pain Manag Nurs. 2015 Feb;16(1):33-9. doi: 10.1016/j.pmn.2014.03.003. Epub 2014 Jun 7. PMID 24912740
- [Background] Shilpapriya M, Jayanthi M, Reddy VN, Sakthivel R, Selvaraju G, Vijayakumar P. Effectiveness of new vibration delivery system on pain associated with injection of local anesthesia in children. J Indian Soc Pedod Prev Dent. 2015 Jul-Sep;33(3):173-6. doi: 10.4103/0970-4388.160343. PMID 26156269